CLINICAL TRIAL: NCT05269680
Title: STAR-LIFE: a Post-market Registry on MINIject
Acronym: STAR-LIFE
Status: Recruiting | Type: Observational
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: STAR-LIFE (ISM11)
Record Dates: First submitted 2022-02-08; First posted 2022-03-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Open Angle Glaucoma
Keywords: Open Angle Glaucoma; Minimally Invasive Glaucoma Surgery; MINIject
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As part of the post-market clinical follow-up (PMCF), this registry is developed to ensure real-world data collection on MINIject device.

DETAILED DESCRIPTION:
The goal of the registry is to collect data of the MINIject in a real-life setting. The registry has 3 main objectives: the collection of real-world evidence on the usability of the device, the patient reported outcomes, and the device safety over a period of 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years
* diagnosed with open angle glaucoma, who has been or will be implanted with CE-marked MINIject
* able to give consent

Exclusion Criteria:

* eyes with angle closure glaucoma
* eyes with traumatic, malignant, uveitic or neovascular glaucoma or discernible congenital anomalies of the anterior chamber angle
* patients with known intolerance or hypersensitivity to silicone
* patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient diagnosed with open angle glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
QoL | 2 years after surgery
  quality of life will be quantified by use of a standardized quality of life questionnaires SHPC-18
ease of use | 1 day
  the usability of the device will be defined by use of a surgeon questionnaire.
Number of participants with treatment-related incidents | up to 2 years after surgery (study completion)
  collection of incidences (nature (ocular or non-ocular), number and severity) throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Universitatsklinik fur Augenheilkunde Inselspital, Bern, Switzerland